CLINICAL TRIAL: NCT05764187
Title: Incidence of White Spot Lesions Around Ceramic Brackets Compared With Metal Brackets Evaluated With Quantitative Light-induced Fluorescence: A Randomized Clinical Trial
Brief Title: Incidence of White Spot Lesions Around Ceramic Brackets Compared With Metal Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: JUST20220107
Record Dates: First submitted 2023-02-04; First posted 2023-03-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: White Spot Lesion of Tooth

STUDY DESIGN:
Intervention Model Description: Two parallel arm randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: It was not possible to mask nether the participants nor the care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ceramic orthodontic brackets (Experimental): Patients bonded with ceramic brackets for orthodontic treatment
  Interventions: Other: Orthodontic fixed appliance therapy
- Metal orthodontic brackets (Active Comparator): Patients bonded with metal brackets for orthodontic treatment
  Interventions: Other: Orthodontic fixed appliance therapy

INTERVENTIONS:
Other: Orthodontic fixed appliance therapy — Follow up of white spot lesion development using quantitative light induced fluorescence in patients bonded with ceramic brackets versus patients bonded with conventional metal brackets

SUMMARY:
The main objective of this study was to investigate the relation between ceramic brackets and the development of white spot lesions (WSLs) compared to that associated with conventional metal brackets.

DETAILED DESCRIPTION:
Objectives : The main objective of this study was to investigate the relation between ceramic brackets and the development of WSL compared to that associated with conventional metal brackets.

Study design: Randomized 2-parallel arm clinical trial. Materials and methods: Quantitative light induced fluorescence (QLF) images were taken for the two randomly allocated groups (Ceramic group, n=26; Metal group, n=25) of patients at T0: before the start of treatment; T1: after 2 months and T2: at 4 months after treatment). The QLF images were analyzed; Primary outcome measures: The lesion area (Pixels) and Mean amount of fluorescence loss (∆F)% and the number of newly developed lesions. Secondary outcome: Maximum fluorescence loss (∆F-Max)% and plaque surface area (∆R 30)%. Means and standard deviations for all the measured parameters at T0, T1 and T2 were calculated. Split plot analysis of variance (SPANOVA) test was used to determine the changes within each group at the different time intervals, and between the two groups. Chi square was used to compare between the two groups regarding the number of new lesions during the treatment. P value was set at 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects seeking orthodontic treatment with mild-to-moderate crowding (not exceeding 5 mm)
* No previous orthodontic treatment
* Optimum oral hygiene
* Maximum of 3 restored teeth
* Absence of defective enamel formation in the form of hypocalcification or hypoplasia.

Exclusion Criteria:

* Subjects with poor oral hygiene
* Defective enamel
* Patients with syndromes and Oro-facial anomalies or salivary glands diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Lesion area | 4 months
  Surface area of the lesion measured in Pixels
Mean fluorescence loss ∆F(%) | 4 months
  Mean lesion fluorescence loss reflecting mineral loss measured in percent
Maximum fluorescence loss ∆Fmax(%) | 4 months
  Deepest point of the lesion
Incidence of white spot lesions | 4 months
  The number of newly developed white spot lesions

SECONDARY OUTCOMES:
Plaque measurement | 4 months
  Amount of plaque around the orthodontic fixed appliance

CONTACTS AND LOCATIONS:
Overall Officials: Susan Al-Khateeb, Professor, Principal Investigator — Faculty of Dentistry/Jordan University of Science and Technology
Locations (1):
- Postgraduate Teaching Dental Clinics/JUST, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request

REFERENCES:
- [Background] Chalmers JM. Minimal intervention dentistry: part 1. Strategies for addressing the new caries challenge in older patients. J Can Dent Assoc. 2006 Jun;72(5):427-33. PMID 16772067
- [Background] Chapman JA, Roberts WE, Eckert GJ, Kula KS, Gonzalez-Cabezas C. Risk factors for incidence and severity of white spot lesions during treatment with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):188-94. doi: 10.1016/j.ajodo.2008.10.019. PMID 20691360
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Birnie D. Ceramic brackets. Br J Orthod. 1990 Feb;17(1):71-4. doi: 10.1179/bjo.17.1.71. PMID 2178681
- [Background] Russell JS. Aesthetic orthodontic brackets. J Orthod. 2005 Jun;32(2):146-63. doi: 10.1179/146531205225021024. PMID 15994990
- [Background] Fournier A, Payant L, Bouclin R. Adherence of Streptococcus mutans to orthodontic brackets. Am J Orthod Dentofacial Orthop. 1998 Oct;114(4):414-7. doi: 10.1016/s0889-5406(98)70186-6. PMID 9790325
- [Background] Rammohan SN, Juvvadi SR, Gandikota CS, Challa P, Manne R, Mathur A. Adherence of Streptococcus mutans and Candida albicans to different bracket materials. J Pharm Bioallied Sci. 2012 Aug;4(Suppl 2):S212-6. doi: 10.4103/0975-7406.100206. PMID 23066254
- [Background] Passariello C, Gigola P. Adhesion and biofilm formation by oral streptococci on different commercial brackets. Eur J Paediatr Dent. 2013 Jun;14(2):125-30. PMID 23758462
- [Background] Raju, A.S., Hegde, N.A., Reddy, V.P., Chandrashekar, B.S., Mahendra, S. and Harishkoushik, S.R. (2013) An in vivo study on bacterial colonization with metal, ceramic and self-ligating brackets: A scanning electron microscopy study. Journal of Indian Orthodontic Society, 47, 88-96.
- [Background] al-Khateeb S, Oliveby A, de Josselin de Jong E, Angmar-Mansson B. Laser fluorescence quantification of remineralisation in situ of incipient enamel lesions: influence of fluoride supplements. Caries Res. 1997;31(2):132-40. doi: 10.1159/000262388. PMID 9118185
- [Background] Al-Khateeb S, Forsberg CM, de Josselin de Jong E, Angmar-Mansson B. A longitudinal laser fluorescence study of white spot lesions in orthodontic patients. Am J Orthod Dentofacial Orthop. 1998 Jun;113(6):595-602. doi: 10.1016/s0889-5406(98)70218-5. PMID 9637561
- [Background] van der Veen MH, de Josselin de Jong E. Application of quantitative light-induced fluorescence for assessing early caries lesions. Monogr Oral Sci. 2000;17:144-62. doi: 10.1159/000061639. PMID 10949838
- [Background] Benson PE, Parkin N, Millett DT, Dyer FE, Vine S, Shah A. Fluorides for the prevention of white spots on teeth during fixed brace treatment. Cochrane Database Syst Rev. 2004;(3):CD003809. doi: 10.1002/14651858.CD003809.pub2. PMID 15266503
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432
- [Background] Houston WJ. The analysis of errors in orthodontic measurements. Am J Orthod. 1983 May;83(5):382-90. doi: 10.1016/0002-9416(83)90322-6. PMID 6573846
- [Background] Park SH, Kim K, Cho S, Chung DH, Ahn SJ. Variation in adhesion of Streptococcus mutans and Porphyromonas gingivalis in saliva-derived biofilms on raw materials of orthodontic brackets. Korean J Orthod. 2022 Jul 25;52(4):278-286. doi: 10.4041/kjod21.283. Epub 2022 Jun 9. PMID 35678009
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] Almosa NA, Sibai BS, Rejjal OA, Alqahtani N. Enamel demineralization around metal and ceramic brackets: an in vitro study. Clin Cosmet Investig Dent. 2019 Feb 28;11:37-43. doi: 10.2147/CCIDE.S190893. eCollection 2019. PMID 30881139
- [Background] Abu Alhaija ES, Al-Khateeb SN, Al-Nimri KS. Prevalence of malocclusion in 13-15 year-old North Jordanian school children. Community Dent Health. 2005 Dec;22(4):266-71. PMID 16379166
- [Background] Lim HW, Park JH, Park HH, Lee SJ. Time series analysis of patients seeking orthodontic treatment at Seoul National University Dental Hospital over the past decade. Korean J Orthod. 2017 Sep;47(5):298-305. doi: 10.4041/kjod.2017.47.5.298. Epub 2017 Jul 27. PMID 28861391
- [Background] O'Reilly MM, Featherstone JD. Demineralization and remineralization around orthodontic appliances: an in vivo study. Am J Orthod Dentofacial Orthop. 1987 Jul;92(1):33-40. doi: 10.1016/0889-5406(87)90293-9. PMID 3300270
- [Background] Holmen L, Thylstrup A, Artun J. Surface changes during the arrest of active enamel carious lesions in vivo. A scanning electron microscope study. Acta Odontol Scand. 1987 Dec;45(6):383-90. doi: 10.3109/00016358709096362. PMID 3481156
- [Background] Ogaard B, Rolla G, Arends J. Orthodontic appliances and enamel demineralization. Part 1. Lesion development. Am J Orthod Dentofacial Orthop. 1988 Jul;94(1):68-73. doi: 10.1016/0889-5406(88)90453-2. PMID 3164585
- [Background] Julien KC, Buschang PH, Campbell PM. Prevalence of white spot lesion formation during orthodontic treatment. Angle Orthod. 2013 Jul;83(4):641-7. doi: 10.2319/071712-584.1. Epub 2013 Jan 4. PMID 23289733
- [Background] Sundararaj D, Venkatachalapathy S, Tandon A, Pereira A. Critical evaluation of incidence and prevalence of white spot lesions during fixed orthodontic appliance treatment: A meta-analysis. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):433-9. doi: 10.4103/2231-0762.167719. PMID 26759794
- [Background] Lucchese A, Gherlone E. Prevalence of white-spot lesions before and during orthodontic treatment with fixed appliances. Eur J Orthod. 2013 Oct;35(5):664-8. doi: 10.1093/ejo/cjs070. Epub 2012 Oct 8. PMID 23045306
- [Background] Al-Anezi SA, Harradine NW. Quantifying plaque during orthodontic treatment: Angle Orthod. 2012 Jul;82(4):748-53. doi: 10.2319/050111-312.1. Epub 2011 Nov 1. PMID 22044115
- [Background] Beberhold K, Sachse-Kulp A, Schwestka-Polly R, Hornecker E, Ziebolz D. The Orthodontic Plaque Index: an oral hygiene index for patients with multibracket appliances. Orthodontics (Chic.). 2012;13(1):94-9. PMID 22567620
- [Background] Freitas AO, Marquezan M, Nojima Mda C, Alviano DS, Maia LC. The influence of orthodontic fixed appliances on the oral microbiota: a systematic review. Dental Press J Orthod. 2014 Mar-Apr;19(2):46-55. doi: 10.1590/2176-9451.19.2.046-055.oar. PMID 24945514